CLINICAL TRIAL: NCT07145541
Title: A Prospective, Interventional Study Assessing the Effectiveness of the AION BIOSYSTEMS, INC. TempShield ("Shield") for Continuous Temperature Monitoring Device in the Pediatric Emergency Depart
Brief Title: AION BIOSYSTEMS, INC. Tempshield for Continuous Tempreature Monitoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AION Biosystems (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00000455
Record Dates: First submitted 2025-07-28; First posted 2025-08-28 (Actual); Results first posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Fever; Sepsis
MeSH Terms: conditions — Fever; Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Aion Tempshield Device (Experimental)
  Interventions: Device: Aion Tempshield Device

INTERVENTIONS:
Device: Aion Tempshield Device — The AION BIOSYSTEMS, INC. tempshield is a skin-applied, continuous temperature monitor. It is battery powered, communicates using Bluetooth LE to a smartphone, then to a clinician dashboard, and is designed to be worn continuously for up to 60 days. Its primary use is for patient monitoring in hospital or post-discharge from a healthcare facility. Through the tempshield system, clinicians can be notified if a patient's temperature exceeds a given threshold. The tempshield system is centered around a non-invasive temperature sensor placed against the patient's skin, in the pectoral region just below the collar bone. The temperature sensor is held in place with a silicone adhesive tape similar to a custom shaped piece of medical tape. The silicone adhesive tape is hypoallergenic.

SUMMARY:
The purpose of this research study is to evaluate the effectiveness of the AION BIOSYTEMS, INC. tempshield ("Shield") temperature monitoring device and platform in detecting body temperature for children 2-4 years old. The ED Research team will be deploying this device on all qualified patients who are awaiting inpatient admission from the emergency department and who have consented to participating in the study. Patients will be asked to keep the device on for a maximum of 7 hours during their stay in the emergency department. There is a potential clinical benefit that fevers will be detected earlier in subjects wearing the AION BIOSTYEMS, INC. tempshield. It is hoped that information gained from the study will help assist clinical care workflow and the treatment of future patients.

DETAILED DESCRIPTION:
A prospective, single site, interventional study assessing the effectiveness for use of the non-invasive wireless temperature monitoring device and platform in detecting body temperature of young children during 1st 7 hours of their stay in the emergency department for patients, between 2-4 years of age. The AION BIOSYSTEMS, INC. tempshield is a skin-applied, continuous temperature monitor. It is battery powered, communicates using Bluetooth LE to a smartphone, then to a clinician dashboard, and is designed to be worn continuously for up to 60 days. Its primary use is for patient monitoring in hospital or post-discharge from a healthcare facility. This study is designed as prospective, interventional study assessing the effectiveness of the AION BIOSYSTEMS, INC. tempshield ("Shield") for continuous temperature monitoring device in the Pediatric Emergency Department. Upon inpatient admission decision entry to the emergency department, a Children's National study staff will be approached for interest and presented with the project and all relevant study materials/documents.Through the tempshield system, clinicians can be notified if a patient's temperature exceeds a given threshold.

The tempshield system is centered around a non-invasive temperature sensor placed against the patient's skin, in the pectoral region just below the collar bone. The temperature sensor is held in place with a silicone adhesive tape similar to a custom shaped piece of medical tape. The silicone adhesive tape is hypoallergenic. Once enrolled, the tempshield wearable device will be placed on the upper chest with gentle, silicon adhesive tape. Study staff will ensure that the device is stable on the subject's chest. In the case that the device will not successfully adhere to the patient's chest, the research team will forego the enrollment of that specific subject due to lack of feasibility. The research team will register the wearable device and connect it to the AION BIOSYSTEMS, INC. Shield app via the Samsung A13. A Samsung phone will be kept in the patient's room to track the tempreature from the device. This phone is used for recording the Oral temperatures taken by the study staff.

Upon activation of the tempshield, participants will be given 60 minutes for the tempshield to acclimate to the environment before an oral temperature measurement is taken. The oral temperature will be taken by the research team using a Welch Allyn 901053 Oral Thermometer and input information into the AION BIOSYSTEMS, INC. app. After the acclimation period, the first measurement of oral temperature using the Welch Allyn oral thermometer will be recorded in the AION BIOSYSTEMS, INC. Shield app by the research team. Following this, measurements of the tempshield sensor temperature will be recorded in the AION BIOSYSTEMS, INC. Shield app 1 ±5 minutes apart. Research coordinators will measure oral temperatures every 2 hours ±1 hour for up to a 24hour period, with a maximum of 6 recordings per pt.. A patient's participation will end once they are discharged from the ED or after 7 hours, whichever comes first. If the patient is moved to in-patient unit, the research coordinator will remove the device from the participant. After 7 hours or at the time of ED discharge, the device will be removed from the participant. If there is no height listed in the EMR, research staff will measure participant height.

In addition to collecting oral temperature every 2 hours, research staff will also recheck placement of AION BIOSYSTEMS, INC. device in adhesive to ensure that the device is still stable in place. If adhesive is not stable, research staff will replace the adhesive with new strip. Research staff will check with LAR to make sure that device was not removed or did not fall off. If device was removed or had fallen off, research team will document estimated time of removal and replacement on CRF and the reasoning for the device displacement. If the device is damage and unable to be used, , the device will be replaced, and the enrollment will continue for the duration of the 7 hours. Otherwise, the same device will be used on the subject throughout the enrollment even if it falls off or is removed from the subject.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients between ages 1 years - 4 years of age
* Confirmed oral temperature of >=99.5 F for febrile participants
* Willing and likely (based on the investigator's judgement) to comply with all study requirements

Exclusion Criteria:

* Participants who are allergic to silicone
* Adolescents with sensory issues who may find it difficult to have a wearable device on their chest.
* Participants presenting an anatomical limitation that would prevent the use of the wearable device

Ages: 1 Year to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2024-01-31 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2024-10-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital, Washington D.C., District of Columbia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred at Children's National Hospital from 1/31/2024 until 9/17/2024.
Period: Overall Study
Arm/Group | AION TempShield Device
Started | 72
Completed | 39
Not Completed | 33

BASELINE CHARACTERISTICS:
Population: 14 participants did not have baseline measures and were lost to follow up
Arm/Group | AION TempShield Device
Number analyzed (Participants) | 58
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 33
Age, Customized [Count of Participants; unit: Participants]
  Age = 2 years | 6
  Age = 3 years | 16
  Age = 4 years | 37
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Difference in Temperature Reported by the AION Tempshield Compared to the Welch Allyn 901053 Electronic Thermometer
Description: Temperature from the study participants will be collected via the AION TempShield and the Welch Allyn 901053 electronic thermometer. The difference output measure was then calculated by subtracting the TempShield-reported temperature from the Welch Allyn temperature.
  I.e., outcome measure = Welch Allyn temperature - TempShield temperature
Time Frame: 24 Hours
Population: 33 participants did not complete the study
Measure: Mean (95% Confidence Interval); unit: degrees Celsius
Arm/Group | AION TempShield Device
Number analyzed (Participants) | 39
degrees Celsius | 0.0 [-0.7 to 0.7]

ADVERSE EVENTS:
Time Frame: From enrollment until ED discharge or device removal, up to 7 hours
Arm/Group | AION TempShield Device
All-Cause Mortality (participants affected / at risk) | 0/72
Serious Adverse Events (participants affected / at risk) | 0/72
Other Adverse Events (participants affected / at risk) | 0/72

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-05-01): https://cdn.clinicaltrials.gov/large-docs/41/NCT07145541/Prot_SAP_000.pdf
  • Informed Consent Form (2024-05-02): https://cdn.clinicaltrials.gov/large-docs/41/NCT07145541/ICF_001.pdf